CLINICAL TRIAL: NCT03056508
Title: Nutrition, Exercise and Lifestyle: Team 6 of the Canadian Consortium on Neurodegeneration in Aging (CCNA)
Brief Title: Lifestyle, Exercise and Diet: The LEAD Study
Acronym: LEAD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19, recruitment and enrollment was suspended and never resumed. COVID-related changes have been made to the clinical program which houses our intervention, and we could not compare new participants with our previous cohort.
Sponsor: Rotman Research Institute at Baycrest (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); Toronto Rehabilitation Institute (Other); The Centre for Memory and Aging (Unknown); University of Waterloo (Other)
Responsible Party: Principal Investigator, Carol Greenwood, Senior Scientist, Rotman Research Institute at Baycrest
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CCNA-NELT
Record Dates: First submitted 2017-02-09; First posted 2017-02-17 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Subjective Cognitive Decline; Age-Related Cognitive Decline
Keywords: diet; nutrition; aerobic exercise; cognition; grey matter; cerebral blood flow; neural activity; resting state connectivity
MeSH Terms: interventions — Exercise; Nutritional Status

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise plus Nutrition (Experimental): 6 months of supervised group exercise plus education and strategy training to alter diet to be consistent with recommendations outlined in our brain health food guide (BHFG).
  Interventions: Behavioral: Exercise plus nutrition
- Exercise (Active Comparator): Identical exercise to the experimental plus education and passive discussion about brain health and healthy lifestyle to control for experimental group nutrition sessions.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise plus nutrition — On the same day as the exercise class, participants will also receive nutrition support. Participants will alter their overall diet to be consistent with recommendations outlined in our brain health food guide (BHFG) and receive diet counseling and strategy training to promote retention and enable this dietary change. For the first two months, diet group sessions will be held on a weekly basis. For the remaining four months, sessions will be divided between group sessions and individual meetings with study dietitians, on a predefined schedule. Participants will submit weekly logs outlining diet goals, plans, successes and obstacles to help direct identification of sequential goals.
  Arms: Exercise plus Nutrition
Behavioral: Exercise — Supervised group exercise will be performed once per week (60 minutes) and self-directed exercise (4 additional aerobic and 2-3 resistance training sessions per week) will be monitored by an exercise diary. The initial walking prescription will be set at ~1.6 km and an intensity equivalent to the anaerobic threshold and/or 60% VO2-peak. Progressions will be made every 2 weeks, increasing distance to a maximum of 6.4 km and then increasing to a max intensity of 80% of VO2-peak and/or max duration of 60 minutes. Heart rate and perceived exertion will be monitored. The program will last 6 months.
  Arms: Exercise

SUMMARY:
This study will explore the impact of an exercise and nutrition (EX+NUTR) , relative to exercise alone (EX) intervention, on brain structure and function as well as blood biomarkers in older adults with subjective cognitive decline (SCD) and vascular risk factors. The overall hypotheses are that a combined EX+NUTR, relative to EX, intervention will evoke more positive changes in brain structure (e.g. hippocampal volume), neural activity (e.g. task associated functional activations monitored through fMRI), and cognitive performance. These changes will be associated with an improved metabolic profile, reductions in inflammatory cytokines and oxidative burden, and greater intervention compliance.

DETAILED DESCRIPTION:
All participants will engage in group supervised exercise sessions once per week as well as engage in additional exercise sessions at home 4 days/week. The exercise program will be run out of two sites (Toronto Rehabilitation Institute (TRI) - Rumsey Centre in Toronto, and the Centre for Community, Clinical Applied Research Excellence (CCCARE) at the University of Waterloo). The supervised exercise sessions modeled after the standard TRI Cardiovascular Prevention and Rehabilitation program, including aerobic training, resistance training and education/counseling. The active group will receive strategy training to simultaneously improve their diet in conjunction with our newly developed Brain Health Food Guide (EX+BHFG); the placebo control group (EX+BHEd) will receive brain health education to control for time and social participation. [NOTE All participants must also be enrolled in the SCD cohort of the CCNA and undergo the CCNA's COMPASS-ND assessment at the beginning of the trial.] The study is 6 months in duration and requires participants to attend 2.5 hr weekly sessions (1 hr supervised exercise, 0.5 hr exercise/stress education and 1 hr nutrition or brain health education) and to exercise on their own an additional 3-4 times per week. Participants are assessed on measures of cognition, brain health (MRI), functional status at baseline, post intervention and 6 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* meeting criteria for subjective cognitive impairment (1 through 5 below)

  1. Answer Yes to both following questions:

     1. Do you feel like your memory or thinking is becoming worse?
     2. Does this concern you?
  2. Have a delayed recall score on 1 paragraph of the Logical Memory test (Wechsler Memory Scale, maximum score 25) above the education-adjusted cut-offs:

     * ≥9 for 16+ years of education;
     * ≥5 for 8-15 years of education;
     * ≥3 for 0-7 years of education.
  3. Have a Montreal Cognitive Assessment (MoCA) total score of 20 and over (≥20/30).
  4. Have a delayed recall score on the CERAD word list of 5 and over (≥5).
  5. Have a global Clinical Dementia Rating score (CDR) equal to 0.5 or less (≤0.5).
* ≥2 vascular risk factors (overweight (BMI>25), T2DM, hypercholesterolemia or hypertension),
* Consuming a poor quality diet (at least median or below on number of servings of vegetable, fruit, fish and nuts based on Canadian consumption patterns in older adults)
* Reasonably sedentary (less than 75min per week of moderate - vigorous intensity physical activity)
* Be available for the whole intervention (6 months) and a 12- month follow-up visit
* English speaking

Exclusion Criteria:

* The presence of significant known chronic brain disease such as: moderate to severe chronic static leukoencephalopathy (including previous traumatic injury), multiple sclerosis, a serious developmental handicap, malignant tumors, Parkinson's disease, and other rarer brain illnesses.
* Ongoing alcohol or drug abuse that in the opinion of the investigator may interfere with the subject's ability to comply with the study procedures.
* Subject does not have a study partner who can provide corroborative information.
* Symptomatic stroke within the previous year.
* Unable to undergo MRI scan due to medical contraindications or inability to tolerate the procedure.
* Major surgery within last 2 months.
* History of intracranial surgery
* Serious comorbid condition that, in the opinion of the study investigator, is likely to result in death within a year.
* High performance athletes

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2020-10-08 (Actual)

PRIMARY OUTCOMES:
Changes from baseline brain structure at 6 months and 12 months. | 6 months plus 6 month follow-up
  Cortical and subcortical grey matter density using MRI three-dimensional T1 weighted structural scan (MPRAGE)

SECONDARY OUTCOMES:
Changes from baseline cerebral blood flow at 6 months and 12 months. | 6 months plus 6 month follow-up
  Pseudo-continuous arterial spin labeling MRI (pcASL) to quantify cerebral blood flow
Changes from baseline cognition at 6 months and 12 months | 6 months plus 6 month follow-up
  pen and paper and computerized tasks, monitoring memory, executive function, and speed of processing. The results will be presented as a composite score of total neuro-psychological performance aggregating scores from the above cognitive domains.
Changes from baseline brain activity related to attention at 6 months and 12 months | 6 months plus 6 month follow-up
  BOLD functional MRI while participants performing an attention task
Changes from baseline resting state connectivity at 6 months and 12 months | 6 months plus 6 month follow-up
  BOLD functional MRI while participants at rest
Changes from baseline diet quality at 6 months and 12 months | 6 months plus 6 month follow-up
  Principle component analyses based on Canadian Diet History Questionnaire II (C-DHQII)
Changes from baseline adherence to diet recommendations at 6 months and 12 months | 6 months plus 6 month follow-up
  Principle component analyses based on the Eating Pattern Self-Assessment
Changes from baseline grip strength at 6 months and 12 months | 6 months plus 6 month follow-up
  Grip strength using a hand held dynamometer
Changes from baseline gait performance at 6 months and 12 months | 6 months plus 6 month follow-up
  Gait velocity, stride length/width, and associated variability assessed using a GAITRite pressure sensor mat.
Changes from baseline balance performance at 6 months and 12 months | 6 months plus 6 month follow-up
  Posturography assessment on balance platform
Changes from baseline maximal oxygen uptake at 6 months and 12 months | 6 months plus 6 month follow-up
  VO2max determined during cardiopulmonary assessment
Changes from baseline blood moderators at 6 months and 12 months | 6 months plus 6 month follow-up
  e.g. BDNF, pro-BDNF, ApoE,
Changes from baseline HbA1C at 6 months and 12 months | 6 months plus 6 month follow-up
  HbA1C
Changes from baseline fasting glucose at 6 months and 12 months | 6 months plus 6 month follow-up
  fasting glucose
Changes from baseline insulin levels at 6 months and 12 months | 6 months plus 6 month follow-up
  insulin
Changes from baseline lipid levels at 6 months and 12 months | 6 months plus 6 month follow-up
  lipid profile
Changes from baseline homocysteine levels at 6 months and 12 months | 6 months plus 6 month follow-up
  homocysteine
Changes from baseline C reactive protein levels at 6 months and 12 months | 6 months plus 6 month follow-up
  CRP
Changes from baseline TNF-alpha levels at 6 months and 12 months | 6 months plus 6 month follow-up
  TNF-alpha
Changes from baseline IL6 levels at 6 months and 12 months | 6 months plus 6 month follow-up
  IL6
Changes from baseline vitamin K levels at 6 months and 12 months | 6 months plus 6 month follow-up
  Vitamin K

CONTACTS AND LOCATIONS:
Overall Officials: Carol E Greenwood, PhD, Principal Investigator — Rotman Research Institute Baycrest Health Sciences; Nicole D Anderson, PhD, Principal Investigator — Rotman Research Institute Baycrest Health Sciences
Locations (4):
- Canada (4):
  - Toronto Rehabilitation Institute Rumsey Centre, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Rotman Research Institute, Toronto, Ontario
  - Centre for Community, Clinical Applied Research Excellence (CCCARE) at the University of Waterloo, Waterloo, Ontario

IPD SHARING:
Plan to Share IPD: Yes
data will be uploaded to shared CCNA database - LORIS

REFERENCES:
- [Derived] Koblinsky ND, Anderson ND, Ajwani F, Parrott MD, Dawson D, Marzolini S, Oh P, MacIntosh B, Middleton L, Ferland G, Greenwood CE. Feasibility and preliminary efficacy of the LEAD trial: a cluster randomized controlled lifestyle intervention to improve hippocampal volume in older adults at-risk for dementia. Pilot Feasibility Stud. 2022 Feb 9;8(1):37. doi: 10.1186/s40814-022-00977-6. PMID 35139918